CLINICAL TRIAL: NCT00952211
Title: Burden of Obstructive Sleep Apnea in Stroke (BOSAST)
Acronym: BOSAST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: problems with recruitment
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Joel E. Dimsdale, M.D., Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HL091848
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Stroke; Obstructive Sleep Apnea
Keywords: stroke; obstructive sleep apnea; fatigue; quality of life
MeSH Terms: conditions — Stroke; Sleep Apnea, Obstructive; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP (Active Comparator): CPAP at therapeutic pressure
  Interventions: Device: CPAP
- sub-therapeutic CPAP (Sham Comparator): CPAP administered at sub-therapeutic pressure
  Interventions: Device: CPAP at sub-therapeutic pressure

INTERVENTIONS:
Device: CPAP — CPAP at therapeutic pressure during nighttime
  Arms: CPAP
Device: CPAP at sub-therapeutic pressure — CPAP delivered at sub-therapeutic pressure at nighttime
  Arms: sub-therapeutic CPAP

SUMMARY:
There are two purposes of this study. The first purpose is to define the frequency of obstructive sleep apnea in stroke survivors as well as its association with fatigue and quality of life. The second purpose is to determine if continuous positive airways pressure (CPAP) treatment can have a beneficial effect on these patients' fatigue and quality of life.

DETAILED DESCRIPTION:
Stroke survivors frequently complain of fatigue, depressive symptoms, and decreased cognitive functioning. These burdens complicate the recovery and rehabilitation from stroke. While there may be many contributing factors to these burdens, one factor in particular may be both terribly common and yet readily susceptible to intervention. Consistent reports from around the world demonstrate that >50% of stroke patients have obstructive sleep apnea (OSA), a disorder that is also associated with fatigue, depressive symptoms, and decreased cognitive functioning. OSA is also associated with increases in inflammatory products which themselves are associated with the same array of burdens.

This study will examine inpatients at a stroke rehabilitation center. Patients' sleep will be studied. Patients with OSA will be randomized to 10 days treatment double blind with either continuous positive airways pressure (CPAP) treatment or to sub-therapeutic CPAP treatment. After 10 days of treatment, the OSA patients and the stroke patient without OSA will be restudied.

The study will shed light on the impact of OSA on stroke patients' burdens.

ELIGIBILITY:
Inclusion Criteria:

* stroke survivor in stroke rehabilitation unit
* age 45-85
* able to consent
* no prior treatment with CPAP

Exclusion Criteria:

* complex apnea
* known inflammatory disease
* neurological disease precluding patient's ability to consent and cooperate

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Dimsdale, MD, Principal Investigator — UCSD
Locations (1):
- UCSD, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tomfohr LM, Hemmen T, Natarajan L, Ancoli-Israel S, Loredo JS, Heaton RK, Bardwell W, Mills PJ, Lee RR, Dimsdale JE. Continuous positive airway pressure for treatment of obstructive sleep apnea in stroke survivors: what do we really know? Stroke. 2012 Nov;43(11):3118-23. doi: 10.1161/STROKEAHA.112.666248. Epub 2012 Sep 27. No abstract available. PMID 23019248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for enrollment on 9/16/09 at San Diego Rehabilitation Institute. Enrollment was halted in April 2011 and the study terminated due to low recruitment numbers.
Period: Overall Study
Arm/Group | CPAP | Sub-therapeutic CPAP
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPAP | Sub-therapeutic CPAP | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 1 |  | 1
Gender [Number; unit: participants]
  Female | 2 |  | 2
  Male | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Profile of Mood States (POMS) - Fatigue Subscale
Description: POMS fatigue subscale: 7 items; range 0-28; higher score indicates worse symptoms, i.e., more fatigue
Time Frame: 10 days after beginning CPAP treatment
Population: Data only available for 2 subjects; one subject did not provide data for this questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CPAP | Sub-therapeutic CPAP
Number analyzed (Participants) | 2 | 0
units on a scale | 10 (2.83) |

2. Secondary Outcome: Hospital Anxiety and Depression (HADS) Scale -Depression Subscale
Description: HADS depression subscale: 7 items, range 0-21. Higher score indicates worse symptoms
Time Frame: 10 days after beginning CPAP treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CPAP | Sub-therapeutic CPAP
Number analyzed (Participants) | 3 | 0
units on a scale | 8 (5) |

ADVERSE EVENTS:
Arm/Group | CPAP | Sub-therapeutic CPAP
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No